CLINICAL TRIAL: NCT02519634
Title: Super-Mini Percutaneous Nephrolithotomy (SMP) Versus Retrograde Intrarenal Surgery (RIRS) for Symptomatic Lower Pole Renal Calculi of 10-20 mm Size: a Randomized Controlled Trial (IAU-01)
Brief Title: SMP vs RIRS for Symptomatic Lower Pole Renal Calculi of 10-20 mm Size: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice President of the Hospital, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRER(45)2015
Record Dates: First submitted 2015-08-03; First posted 2015-08-11 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Renal Calculi
Keywords: Super-Mini Percutaneous Nephrolithotomy; SMP; Retrograde Intrarenal Surgery; RIRS; Randomized Controlled Trial; RCT
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Patients in Group 1 undergo Super-Mini Percutaneous Nephrolithotomy
  Interventions: Procedure: Super-Mini Percutaneous Nephrolithotomy
- Group 2 (Other): Patients in Group 2 undergo Retrograde Intrarenal Surgery
  Interventions: Procedure: Retrograde Intrarenal Surgery

INTERVENTIONS:
Procedure: Super-Mini Percutaneous Nephrolithotomy — Patients undergo Super-Mini Percutaneous Nephrolithotomy
  Arms: Group 1
Procedure: Retrograde Intrarenal Surgery — Patients undergo Retrograde Intrarenal Surgery
  Arms: Group 2

SUMMARY:
Shock wave lithotripsy (SWL) is recommended for kidney stones < 20 mm. However, the stone clearance of lower pole calculi after SWL is limited, thus leading to an extended indication for mini-percutaneous nephrolithotripsy (PCNL) even for stones between 10 and 20 mm in many centers. This trend is further promoted by introduction of super-mini PCNL (SMP), which is postulated to be less invasive compared to mini-PCNL due to the miniaturized instruments. However, this issue remains controversial.

On the other hand, improvements in endoscopy technology have made retrograde stone removal more attractive. This has led to an increasing use of RIRS as a primary treatment although it is recommended only as 2nd-line option by current guidelines. However, the treatment of symptomatic lower pole calculi is a challenge for RIRS because of lower clearance rates.

The purpose of this study is to evaluate the efficacy and safety of SMP and RIRS for the treatment for symptomatic lower pole calculi renal calculi measuring 10-20 mm.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of SMP and RIRS for the treatment for symptomatic lower pole calculi renal calculi measuring 10-20 mm.Investigators will do a multi-centers international randomized controlled trial(RCT)，and investigators plan to perform this study in 10 hospitals，which are the First Affiliated Hospital of Guangzhou Medical University of China, Department of Urology, Renmin Hospital, Wuhan University of China, Shenzhen People's Hospital of China, The Second Affiliated Hospital of Zhengzhou University of China, The Second Affiliated Hospital of Harbin Medical University of China, Zhujiang Hospital of Southern Medical University of China, Jiangsu Province hospital, The First Affiliated Hospital With Nanjing Medical University of China, Zhejiang provincial people's hospital of china, Dr. Lutfi Kirdar Training and Research Hospital of Turkey and Global Rainbow Healthcare of India respectively.

Investigators plan to beginning their study at August in 2015 and end at July in 2017.One hundred and sixty patients with symptomatic lower pole calculi renal calculi measuring 10-20 mm will be enrolled in this study. By simple random sampling technique, patients will be assigned to two 80-patient groups.All the patients will be diagnosed definitely before operations with non-contrast CT.Patients with positive preoperative urine culture should be treated with suitable antibiotics based on the culture sensitivity result for at least 72h before SMP/RIRS. Patients who have negative urine culture should receive a single dose of broad spectrum antibiotic prophylaxis just prior to the procedure.

Surgical technique

SMP

All the biochemistry tests and preoperative preparations are referenced to the mini-PCNL. Under general anesthesia a 6 French(Fr).Open end ureteral catheter is first inserted in to the relevant ureter. Patient is then turned into prone position and the desired calyx is punctured under fluoroscopic or sonographic guidance. Nephrostomy tract dilation is carried out using fascial dilators up to 12-14 Fr. as indicated. Corresponding size of suction-evacuation sheath was placed. The sheath is connected to the specimen collection bottle and the bottle then onto the aspirator. A rubber cap with a center aperture was placed at the proximal end of the sheath. The negative pressure aspirator was adjusted to a setting of 150-200 mm Hg. The miniature endoscope is inserted into the sheath through the cap. Stone is visualized and lithotripsy is performed using either Holmium-yttrium aluminum garnet(YAG) laser or pneumatic lithotripsy. At the end of procedure fluoroscopic images are obtained to assess stone clearance status. Double J ureteral stent is placed only in the presence of ureteral inflammatory polyp; evidence of ureteropelvic obstruction; presence of significant pyelocalyceal blood clots following lithotripsy; significant residual stones. Indications for nephrostomy tube placement included: significant residual stone fragments which would require a second look procedure; significant pyelocalyceal blood clots or bleeding after lithotripsy (because the nephrostomy tube could tamponade the access tract and drain the urine and clots).

RIRS

The patient is placed in the lithotomy position, Cystoscopy and retrograde pyelogram were preformed, and a 0.035'' flexible tip guidewire is placed into the renal pelvis. A 12 Fr/ 14 Fr ureteral access sheath (UAS) is advanced into the proximal ureter over the guidewire, and a P5 or P6 Olympus flexible ureteroscope is passed through the UAS. The stones are fragmented using a 200um holmium laser fibre at a 8-25 weeks energy setting. Some fragments are removed using a stone basket for stone analysis, and the remaining stone fragments smaller than 2 mm were left for spontaneous passage. A 5 Fr or 6Fr pigtail stent is placed at the conclusion of the procedure. Double J stents were removed post-operative 2 weeks.

Data collection

Data for the 2 groups-demographic characteristics,hemoglobin(HB) decrease, postoperative pain, duration of postoperative, hospital stay, complications (modified Clavien system), stone clearance (SFR after day 1 and final SFR) and the need for auxiliary treatment are compared.

Mean study endpoint: The primary endpoint was the SFR at 3-months after surgery.

Secondary endpoint: Complications, duration of postoperative and hospital stay. re-SMP, ureteroscopy and SWL are considered as auxiliary treatments. Demographic characteristics include age, sex, BMI, stone size and location, etc…

The stone size is defined as the maximum diameter as determined by CT scans.

Degree of hydronephrosis are assigned as follow: none (no calyx or pelvic dilation), mild (pelvic dilatation alone), moderate (mild calyx dilation), or severe (severe calyx dilation or calyx dilation accompanied by renal parenchyma atrophy).

Definition of operation time:

For SMP: recorded from the time of the first percutaneous renal puncture to the completion of the stone removal.

For RIRS: recorded from insertion of an endoscope into the urethra to the completion of stent placement.

Hospital stay are rounded to the nearest whole day and calculated from the day of surgery to the day of discharge.

Postoperative pain (visual analogue scale(VAS), use of analgesics) and Postoperative comfort scores (Bruggrmann comfort scale，BCS) will be recorded.

The rate of hemoglobin decrease is assessed by comparing the preoperative Hb level with 24-hour postoperative Hb level.

SFR is assessed by KUB and ultrasound at 1-day after operation.

Non-contrast CT is obtained for all patients at 3 month after the operation to evaluate the final SFR, allowing time for the spontaneous passage of stone fragments.

Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were defined as ≦ 3mm, asymptomatic, non-obstructive and non-infectious stone particles.

If the procedure is considered as successful, the pigtail stent is removed as outpatient after 2 weeks. Follow-up including non-contrast CT will be generally scheduled in 3 month.

Bleeding severity is judged by the treating physician, and transfusions are administered according to local practice guideline.

Complications of all patients are recorded according to modified Clavien classification system.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years
2. Normal renal function
3. Anesthesia rating(ASA) score 1 and 2
4. Absence of congenital abnormalities
5. Symptomatic lower pole calculi and diameter 10-20 mm

Exclusion Criteria:

1. Patients with solitary kidney
2. Patients with congenital anomalies, e.g. ectopic kidney, polycystic horseshoe, or mal-rotated kidney
3. Patients who underwent transplant or urinary diversion
4. Uncorrected coagulopathy and active urinary tract infection(UTI)
5. Patient undergoing any other surgical procedure during the same admission. (e.g. ureteroscopy)
6. If patients undergoing RIRS/SMP have purulent urine, we will place D-J stent (for RIRS) or nephrostomy tube (for SMP) and postpone the procedure and excluded the patients from the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Stone free rate (SFR) | The primary endpoint was the SFR at 3-months after surgery.
  Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were defined as ≦ 3mm, asymptomatic, non-obstructive and non-infectious stone particles.

SECONDARY OUTCOMES:
Perioperative complications | intraoperatively or ≤ 3 month postoperatively
  Complication is defined as any adverse event occurred intraoperatively or ≤3 month postoperatively.
Operation time | intraoperatively
  The operating time for SMP was recorded from the time of the first percutaneous renal puncture to wound closure;For RIRS,The operating time was recorded from insertion of an endoscope into the urethra to the completion of stent placement.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Department of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zeng G, Zhang T, Agrawal M, He X, Zhang W, Xiao K, Li H, Li X, Xu C, Yang S, de la Rosette JJ, Fan J, Zhu W, Sarica K. Super-mini percutaneous nephrolithotomy (SMP) vs retrograde intrarenal surgery for the treatment of 1-2 cm lower-pole renal calculi: an international multicentre randomised controlled trial. BJU Int. 2018 Dec;122(6):1034-1040. doi: 10.1111/bju.14427. Epub 2018 Jul 26. PMID 29873874